CLINICAL TRIAL: NCT01765283
Title: A Prospective, Open Label, Multicenter, Partially Randomized, Safety Study of One Cycle of Promethera HepaStem in Urea Cycle Disorders (UCD) and Crigler-Najjar Syndrome (CN) Paediatric Patients.
Brief Title: Safety Study of HepaStem for the Treatment of Urea Cycle Disorders (UCD) and Crigler-Najjar Syndrome (CN)
Acronym: HEP001
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cellaion SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEP001
Record Dates: First submitted 2013-01-09; First posted 2013-01-10 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Urea Cycle Disorders; Crigler Najjar Syndrome
Keywords: CN,; UCD
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Crigler-Najjar Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hepastem Low dose (Experimental): 12.5x106cells/kg
  Interventions: Biological: HepaStem
- Hepastem Intermediate dose (Experimental): 50x106cells/kg
  Interventions: Biological: HepaStem
- Hepastem High dose (Experimental): 200x106cells/kg
  Interventions: Biological: HepaStem

INTERVENTIONS:
Biological: HepaStem
  Other Names: HHALPC,Heterologous Human Adult Liver derived Progenitor Cells

SUMMARY:
The purpose of this study is to assess the safety and to appraise the efficacy of one cycle of Hepastem (Heterologous Human Adult Liver-derived Progenitor Cells, HHALPC) infusions in paediatric patients suffering from CN or UCD.

The study duration: 12 months starting from the day of treatment: 6 months active surveillance and 6 months observation post-infusion.

ELIGIBILITY:
GENERAL:

1. Subject shows patency of the portal vein and branches, with normal flow velocity in the main portal vein as confirmed by Doppler ultrasound and accessibility of the portal vein, or respectively, accessibility of the umbilical vein.
2. Subject (if capable of signing) and parents or legal representative have provided a written informed assent/consent.
3. Female subjects of childbearing potential need to have a negative pregnancy test and must agree to use an acceptable method of contraception throughout the study.

MAIN INCLUSION CRITERIA

Crigler-Najjar Syndrome specific:

* Patient presents with Crigler-Najjar syndrome type 1.
* Patient presents with Crigler-Najjar syndrome type 2, poorly controlled under phenobarbital treatment, or experiencing serious impairment in quality of life.

Diagnosis must be confirmed by genetic mutation analysis if not available.

Urea Cycle Disorders specific:

* Diagnosis of one of the urea cycle disorders of which the disease is of such severity to warrant liver transplantation or alternatives despite full conservative therapy,
* subject experiencing serious impairment in quality of life despite full conservative therapy.

MAIN EXCLUSION CRITERIA

* The subject is 18 years or older at time of screening.
* The subject presents acute liver failure, clinical or radiological evidence of liver fibrosis or cirrhosis, presents or has a history of hepatic or extrahepatic malignancy
* The patient has a non-corrected cardiac malformation, has a known medical or family history of coagulopathy, had or has a renal insufficiency treated by dialysis.
* The subject requires valproate therapy.
* The subject has a thrombosis of the portal vein or persisting impairment of anterograde portal blood flow.
* The subject has a porto systemic shunt or fistula assessed by Doppler US.
* Patients with disease of such severity that liver transplantation is an absolute indication.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2014-10 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Safety of HepaStem in paediatric patients suffering from CN or UCD | 6 months
  Evaluation of the clinical status, portal-vein hemodynamics, morphology of the liver, de novo detection of circulating anti-HLA antibodies, and/or other immune related markers as well as Serious Adverse Events (SAEs) and clinically significant Adverse Events (AEs) related to infusion.

SECONDARY OUTCOMES:
Long-term safety profile of HepaStem in both indications | From 6 to 12 months post-administration
  Assessment of reactogenicity and safety of the treatment during 6 to 12 months post infusion (long-term safety) is evaluated.
Preliminary efficacy of HepaStem in both indications (CN and UCD) and for different weight cohorts | 0-6 months, 6-12 months
  UCD: 13C tracer test to measure ureagenesis, ammonium values, amino acids in plasma, neuropsychological assessment and quality of life indicators: (1) report on actual supportive treatment and any adjustment of diet (protein restriction (low protein diet) and amino acids supplements). (2) report on cognitive skills, behaviour, and health related quality of life effect).
  CN: measure of the blood unconjugated bilirubin and serum total bilirubin levels and quality of life indicators: (1) adjustment of duration of phototherapy, (2) report on cognitive skills, behaviour, and (3) health related quality of life effect.

OTHER OUTCOMES:
To characterize the engraftment of HepaStem | at 6 month, and optional at 12 month.
  By liver biopsy, enzymatic activity (quantitative) on the biopsies or, donor sequences by RT PCR or in situ hybridisation (FISH) or immunohistochemistry.

CONTACTS AND LOCATIONS:
Locations (11):
- Belgium (2):
  - Saint Luc University Hospital, Brussels
  - Universitair Ziekenhuis (UZ) Antwerpen, Edegem
- France (3):
  - CHU Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Jeanne de Flandre, CHRU Lille, Lille
  - Hôpital des Enfants, CHU de Toulouse, Toulouse
- Israel (3):
  - Rambam Medical Center, Meyer Children's Hospital, Haifa
  - Hadassah Ein-Kerem Medical Center, Jerusalem
  - Schneider Children's Medical Center of israel, Petah Tikva
- Ospedale Pediatrico Bambino Gesu di Roma, Roma, Italy
- United Kingdom (2):
  - Birmingham Children's Hospital, Birmingham
  - Great Ormond Street Hospital London, London

REFERENCES:
- [Derived] Coppin LCF, Smets F, Ambroise J, Sokal EEM, Stephenne X. Infusion-related thrombogenesis by liver-derived mesenchymal stem cells controlled by anticoagulant drugs in 11 patients with liver-based metabolic disorders. Stem Cell Res Ther. 2020 Feb 7;11(1):51. doi: 10.1186/s13287-020-1572-7. PMID 32028991